CLINICAL TRIAL: NCT03789006
Title: Efficiency of Antithymocyte Globulin and Azathioprine Versus Basiliximab and Mycophenolate Mofetil When Used in Combination With Tacrolimus and Prednisolone in Living Donor Kidney Transplantation
Brief Title: Antithymocyte Globulin and Azathioprine Versus Basiliximab and Mycophenolate Mofetil in Living Donor Kidney Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Khartoum (Other)
Collaborators: National Center for Kidney Diseases and Surgery (Unknown)
Responsible Party: Principal Investigator, Sarra Elamin, Consultant Physician and Nephrologist, University of Khartoum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 033546
Record Dates: First submitted 2018-12-25; First posted 2018-12-28 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Kidney Transplant Rejection
MeSH Terms: interventions — Antilymphocyte Serum; Basiliximab

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATG (Active Comparator): Induction with antithymocyte immunoglobulin (Rabbit) (Grafalon) and maintenance with tacrolimus, azathioprine and prednisolone
  Interventions: Drug: Antithymocyte Immunoglobulin (Rabbit)
- BAS (Active Comparator): Induction with interleukin 2 receptor antagonist (basiliximab) and maintenance with tacrolimus, mycophenolate mofetil and prednisolone
  Interventions: Drug: Interleukin 2 Receptor Antagonist

INTERVENTIONS:
Drug: Antithymocyte Immunoglobulin (Rabbit) — Induction agent for living donor kidney transplantation
  Other Names: grafalon
  Arms: ATG
Drug: Interleukin 2 Receptor Antagonist — Induction agent for living donor kidney transplantation
  Other Names: Basiliximab
  Arms: BAS

SUMMARY:
Kidney transplantation is the best available treatment option for patients with end stage renal disease. However, kidney transplantation requires life-long use of immunosuppressive medication. Because of the high cost of these medications we need to carefully evaluate the cost-effectiveness of each drug regimen, especially in low-middle income countries. The objective of this clinical trial is to compare the efficiency and cost of two immunosuppressive protocols after living donor kidney transplantation: (1) antithymocyte globulin, tacrolimus, azathioprine and prednisolone versus (2) basiliximab, tacrolimus, mycophenolate mofetil and prednisolone.

ELIGIBILITY:
Inclusion Criteria:

* Adult end-stage renal disease patients
* First living donor kidney transplant.
* Moderate immunological risk.

Exclusion Criteria:

* Low immunological risk (HLA mismatches 000/100/010/110 with negative PRA).
* High immunological risk (child to mother or husband to wife transplant, 2 DR mismatches).

  * Known hypersensitivity to any of the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-03-21 (Actual); Primary Completion 2022-03-21 (Estimated); Study Completion 2024-03-21 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute rejection | 6 months post kidney transplant
  The incidence of acute rejection will include clinically diagnosed and biopsy proven acute rejection. Clinically diagnosed rejection includes at least 30% acute rise in serum creatinine level. Biopsy proven rejection will include both cellular and antibody mediated rejection according to Banff 2017 criteria
One year graft survival | 1 year post kidney transplant
  One year kidney allograft survival, uncensored for patient death

SECONDARY OUTCOMES:
Cost of immunosuppressive medication | 1 year post kidney transplant+
  Overall cost of immunosuppressive medication during first year post kidney transplant

CONTACTS AND LOCATIONS:
Overall Officials: Sarra Elamin, MD, Principal Investigator — Consultant Nephrologist
Locations (1):
- Doctor Salma Center for Kidney Diseases, Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: Undecided